CLINICAL TRIAL: NCT00703092
Title: Pilot Study: Role of Dietary Fiber in PCOS Anovulation
Brief Title: Pilot Study:Role of Dietary Fiber in PCOS Anovulation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: P.I. left University. Study terminated
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM11246; 2U54HD034449 (NIH)
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: PCOS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fiber-Stat (Experimental): 2 tablespoons daily
  Interventions: Drug: Fiber-Stat

INTERVENTIONS:
Drug: Fiber-Stat — Liquid fiber supplement, 2 tablespoons twice daily.

SUMMARY:
The purpose of this study is to determine whether 6 months of fiber supplementation will improve ovulation in women with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
We hypothesize that 6 months of fiber supplementation will improve ovulation in women with PCOS by improving insulin sensitivity independent of weight loss. In this pilot study, we will determine the feasibility of conducting a larger double-blind, randomized trial in women with PCOS to test this hypothesis. We will evaluate 15 women over a 10-month period, starting with a 4-month intervention-free observation period to determine the effect on ovulation of adding up to 22g/day of fiber supplementation to their usual weight-maintenance diets (to achieve 28-36 g fiber/day assuming baseline dietary fiber intake, could feasibly be translated into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS between the ages of 18-45 years and with a body mass index of less than or equal to 45
* Less than or equal to 8 periods annually
* elevated serum free testosterone concentrations
* normal thyroid function tests and serum prolactin
* exclusion of late-onset adrenal hyperplasia
* acceptable health based on interview, medical history,physical examination, and lab tests
* ability to comply with the requirements of the study
* ability and willingness to provide signed, witnessed informed consent

Exclusion Criteria:

* Diabetes mellitus
* Clinically significant pulmonary,cardiac ,renal,hepatic,neurologic,psychiatric,infectious,and malignant disease
* high blood pressure
* current or recent(within 2 months prior to study entry) injection of any drugs known or suspected to affect reproductive function including oral contraceptives,metformin,thiazolidinediones,glucocorticoids, GnRH-agonists, or anti-androgens (spironolactone,flutamide,etc)
* documented or suspected history of use of recent (within one year) illicit drug abuse or alcoholism
* ingestion of any investigational drugs within 4 weeks prior to study onset
* pregnancy or lactation(less than or equal to 6 weeks postpartum)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulina A Essah, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- VCU General Clinical Research Center, Richmond, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.vcu.edu/pcos

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fiber-Stat
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Fiber-Stat
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Generate Preliminary Data on the Range of Outcome Measures at Baseline and After 6 Months of Fiber Supplementation in Terms of: Ovulation Rates, Insulin Sensitivity, Concentrations of Circulating Androgens and Satiety.
Time Frame: 10 months
Population: This study was terminated early due to lack of enrollment. No assays were run so there is no data to report.
Arm/Group | Fiber-Stat
Number analyzed (Participants) | 0

2. Secondary Outcome: Quantify Enrollment Strategies, Retention, Compliance, Participant Characteristics, and Data Collection Challenges.
Time Frame: 10 months
Population: This study was terminated early due to lack of enrollment. No assays were run so there is no data to report.
Arm/Group | Fiber-Stat
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Fiber-Stat
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No